CLINICAL TRIAL: NCT02962869
Title: Human Photoallergy Test
Brief Title: Human Photoallergy Test (824/2016)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 18824
Record Dates: First submitted 2016-11-10; First posted 2016-11-11 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAY987517 (Experimental): All subjects are patched with the same product
  Interventions: Drug: BAY987517; Other: Untreated skin

INTERVENTIONS:
Drug: BAY987517 — 50 μl/ cm*2 of the test article is applied directly to two sites on the skin and covered with the appropriate patch. Twenty-four (24) hours later, the patches are removed. The test sites are lightly wiped with a dry cloth/tissue and 3μl/ cm*2 of test article is reapplied directly to the skin of the test site designated for irradiation, and lightly spread over the test site. Forty-eight (48) hours later the procedure is repeated to the same test sites. This process is repeated twice weekly for a total of six exposures. (Formulation number: Z43-078)
Other: Untreated skin — One site is patched without treatment as control

SUMMARY:
To evaluate the potential of a test material to produce a photoallergic response

ELIGIBILITY:
Inclusion Criteria:

* be male or female between the ages of 18 and 60 inclusive
* be lightly pigmented (Fitzpatrick Skin Type I, II, III)
* have read and signed the written Informed Consent Form and have completed a HIPAA Authorization Form (Health Insurance Portability and Accountability Act) in conformance with 45CFR Parts 160 and 164
* be in general good health as determined by the subject's medical history and in the discretion of the investigator

Exclusion Criteria:

* have a visible sunburn
* have a history of sun hypersensitivity/photosensitivity or photosensitive dermatoses
* have a known hypersensitivity or allergy against any of the active and non-active ingredients of the investigational products
* subjects who are employees of the CRO (Contract Research Organization) and/or Bayer or is a household member of an employee

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Intensity of skin reactions is evaluated by 5 point scale | Up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Piscataway, New Jersey, United States